CLINICAL TRIAL: NCT04525638
Title: A Phase II Single Arm Trial Evaluating the Preliminary Efficacy of the Combination of 177Lu-DOTATATE and Nivolumab in Grade 3 Well-differentiated Neuroendocrine Tumours (NET) or Poorly Differentiated Neuroendocrine Carcinomas (NEC)
Brief Title: A Clinical Study to Assess the Combination of Two Drugs (177Lu-DOTATATE and Nivolumab) in Neuroendocrine Tumours
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación de investigación HM (Other)
Collaborators: Syntax for Science, S.L (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMH008
Record Dates: First submitted 2020-08-21; First posted 2020-08-25 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Neuroendocrine Tumours (NET); Neuroendocrine Carcinomas (NEC)
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoma, Neuroendocrine | interventions — lutetium Lu 177 dotatate; Nivolumab

STUDY DESIGN:
Intervention Model Description: open-label, single-arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 177Lu-DOTATATE + Nivolumab (Experimental): Patients will receive 240 mg flat dose of nivolumab intravenously as a 30-minutes infusion and 7.4 GBq 177Lu-DOTATATE intravenously as a 4-hours infusion
  Interventions: Drug: 177Lu-Dotatate; Drug: Nivolumab

INTERVENTIONS:
Drug: 177Lu-Dotatate — 7.4 GBq 177Lu-DOTATATE intravenously as a 4-hours infusion
Drug: Nivolumab — 240 mg flat dose of nivolumab intravenously as a 30-minutes infusion

SUMMARY:
This is a prospective, multi-centre, open-label, single-arm, stratified, exploratory, Phase 2 study evaluating the efficacy and safety of 177Lu-DOTATATE in combination with nivolumab in adult patients with Grade 3 neuroendocrine tumours (NET) or neuroendocrine carcinomas (NEC).

DETAILED DESCRIPTION:
Patients will have unresectable advanced, recurrent or metastatic, histologically confirmed, well-differentiated Grade 3 NET or poorly-differentiated NEC of the pancreas, gastrointestinal tract lung and unknown primary site. Thirty patients will be included in this trial, of which 15 will not have received prior chemotherapy (Cohort 1) and 15 will have received at least one prior line of chemotherapy (Cohort 2). Patient will receive 240 mg flat dose of nivolumab intravenously as a 30-minutes infusion and 7.4 GBq 177Lu-DOTATATE intravenously as a 4-hours infusion. Nivolumab will be administered at Day 1 and Day 15 of a 28-days cycle, starting on Cycle 1 Day 1. Patients will receive the study drugs while it is considered to be in their best interest, 177Lu-DOTATATE being administered at a maximum of 4 injection cycle. Treatment discontinuation criteria include, among others, progression, unacceptable toxicity or patient study withdrawal

ELIGIBILITY:
Inclusion Criteria:

1. Patients having voluntarily signed and dated IRB/IEC-approved written informed consent form in accordance with regulatory and institutional guidelines before the performance of any protocol-related procedures.
2. Patients with advanced/metastatic, histologically confirmed, well-differentiated Grade 3 NET or poorly-differentiated NEC of the pancreas, gastrointestinal tract, lung and unknown primary site at diagnosis or after progression to one systemic treatment. Patients will be enrolled in two cohorts based on the therapy of their aforementioned cancer: Cohort 1: Patients with no previous chemotherapy. Cohort 2: Patients who have received one line of chemotherapy.
3. Age ≥18 years.
4. Patients must have measurable disease based on RECIST v.1.1 meeting the following criteria:

   1. Lesions that have had external beam radiotherapy or loco-regional therapies such as radiofrequency ablation or liver embolization must show evidence of progressive disease based on RECIST v.1.1 to be deemed a target lesion.
   2. Patients in cohort 2 must show evidence of disease progression by radiologic image techniques according to RECIST v.1.1 within 3 months prior to signing informed consent.
5. Confirmed presence of somatostatin receptors on tumour lesions based on positive PET-Gallium (SomaKit) imaging within 8 weeks prior to enrolment in the study. At least one lesion should have an uptake of 64-Gallium higher than the normal liver according to investigator judgement.
6. Karnofsky Performance Score ≥ 60 and Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2.
7. Life expectancy of ≥ 6 months.
8. Adequate normal organ and marrow function as defined below:

   1. Haemoglobin concentration ≥ 8.0 g/dL (5.0 mmol/L).
   2. WBC ≥ 2x10 9/L (2000/mm3).
   3. Platelets ≥75x10 9/L (75x103/mm3).
9. Adequate renal function defined as serum creatinine ≤150 μmol/L or 1.7 mg/dL, or a creatinine clearance or measured glomerular filtration rate (using plasma clearance methods) of ≥ 50 mL/min.
10. Adequate hepatic function defined as total bilirubin ≤3 x ULN and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN (≤ 5 x ULN if liver metastases are present).
11. Serum albumin ≥ 3.0 g/dL (or serum albumin < 3.0 g/dL if prothrombin time is within the normal range).
12. Female patients must either be of non-reproductive potential (i.e., post-menopausal by history: ≥60 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry. Both women and men must agree to use a medically acceptable method of contraception throughout the treatment period and for six months after discontinuation of treatment. Acceptable methods of contraception include intrauterine device, oral contraceptive, subdermal implant and/or double barrier.
13. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow-up.
14. Recovery to Grade ≤ 1 from any adverse event (AE) derived from previous treatment (excluding alopecia and/or cutaneous toxicity and/or asthenia).

Exclusion Criteria:

1. Treatment with >30 mg Octreotide LAR at 3-4 weeks intervals within 12 weeks prior to enrolment in the study.
2. Peptide receptor radionuclide therapy (PRRT) at any time prior to enrolment in the study.
3. Targeted surgery, radiotherapy (external beam), chemotherapy, embolization, interferons, mTOR-inhibitors or other investigational therapy within 12 weeks prior to enrolment in the study. In Cohort 2, chemotherapy should be administered at least 4 weeks prior to first dose of the treatment.
4. Prior treatment with anti-PDL-1/anti-PD-1 or anti-CTL-4 therapy.
5. Known brain metastases, unless these metastases have been treated and stabilized for at least 24 weeks prior to enrolment in the study. Patients with a history of brain metastases must have a head CT with contrast to document stable disease prior to enrolment in the study.
6. Uncontrolled congestive heart failure (NYHA II-IV).
7. Uncontrolled diabetes mellitus as defined by a fasting blood glucose >2 ULN.
8. Any patient receiving treatment with short-acting Octreotide, which cannot be interrupted for 24 h before and 24 h after the administration of 177Lu-DOTATATE , or any patient receiving treatment with Octreotide LAR, which cannot be interrupted for at least 6 weeks before the administration of 177Lu-DOTATATE, unless the tumour uptake observed by Somakit imaging during continued Octreotide treatment is at least as high as normal liver uptake observed by planar imaging.
9. Acute or chronic hepatitis B (e.g., Hepatitis B surface antigen reactive), hepatitis C (e.g., HCV RNA [qualitative] is detected) or known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
10. Active, known, or suspected autoimmune disease within the past 2 years. NOTE: Patients with Type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) and Grave's disease not requiring systemic treatment within the past 2 years are not excluded.
11. Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of start of study treatment. NOTE: Inhaled or topical steroids, and systemic steroid doses > 10 mg daily prednisone equivalent for adrenal replacement are permitted in the absence of active autoimmune disease.
12. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
13. History of allogeneic organ transplant.
14. Known hypersensitivity to nivolumab, 177Lu-DOTATATE or its excipients.
15. Patients with any other significant medical, psychiatric, or surgical condition, currently uncontrolled by treatment, which may interfere with completion of the study. Patients must have recovered from the effects of major surgery or significant traumatic injury at least 14 days before starting treatment.
16. Prior external beam radiation therapy to more than 25% of the bone marrow.
17. Urinary incontinence.
18. Subjects with previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, esophageal, colon, endometrial, cervical/dysplasia, melanoma, or breast) unless a complete remission was achieved at least 5 years prior to study entry AND no additional therapy is required during the study period
19. Prisoners or patients who are compulsory detained.
20. Established or suspected pregnancy or when pregnancy has not been excluded
21. Kidney failure with creatinine clearance < 30 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-29 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Week 15 (+/-1) of treatment
  ORR assessed by RECIST v.1.1

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Week 31 (+/-1) of treatment
  1. ORR assessed by RECIST v.1.1
  2. ORR assessed by Choi and modified RECIST for immune based therapeutics (iRECIST)
Progression-free Survival (PFS) | Week 31 (+/-1) of treatment
Number and Grade of Adverse Events | Week 31 (+/-1) of treatment
  by CTCAE v.5 criteria
Overall Survival (OS) | Week 31 (+/-1) of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cubillo, MD, Study Director — Director
Locations (5):
- Spain (5):
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela, Galicia
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Madrid Sanchinarro, PAU de Sanchinarro, Madrid
  - Hospital Unviersitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No